CLINICAL TRIAL: NCT07073495
Title: A Prospective Observational Study Comparing Edge Laminar Block (ELB) and Serratus Posterior Superior Intercostal Plane Block (SPSIPB) for Postoperative Pain Management After Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: Comparison of Edge Laminar Block and Serratus Posterior Superior Intercostal Plane Block for Postoperative Pain Management After VATS
Acronym: ELB vs SPSIPB
Status: Recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Eda Cennet Caferoğlu, Dr. Eda Cennet Caferoğlu, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-06/84
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Thoracic Surgery; Video-assisted Thoracoscopic Surgery (VATS); Serratus Posterior Superior Intercostal Plane Block; Edge Laminar Block
Keywords: Edge Laminar Block (ELB); Serratus Posterior Superior Intercostal Plane Block (SPSIPB); Video-Assisted Thoracoscopic Surgery (VATS); Postoperative Pain; Pain Assessment; Thoracic Surgery; Opioid Sparing; Interfascial Plane Blocks
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ELB Group: Patients undergoing VATS who received Edge Laminar Block (ELB) for postoperative pain management. ELB involves the injection of local anesthetic at the edge of the thoracic lamina as a regional anesthesia technique. The efficacy and safety of ELB will be evaluated in this group.
- SPSIPB Group: Patients undergoing VATS who received Serratus Posterior Superior Intercostal Plane Block (SPSIPB) for postoperative pain management. SPSIPB involves the injection of local anesthetic into the intercostal plane beneath the serratus posterior superior muscle. The efficacy and safety of SPSIPB will be evaluated in this group.

SUMMARY:
This prospective observational study aims to compare the effectiveness of Edge Laminar Block (ELB) and Serratus Posterior Superior Intercostal Plane Block (SPSIPB) in managing postoperative pain after Video-Assisted Thoracoscopic Surgery (VATS). The study will evaluate postoperative pain scores (VAS/NRS), opioid consumption, incidence of postoperative nausea and vomiting (PONV), additional analgesic requirements, and patient satisfaction between the two regional analgesic techniques. This research seeks to provide guidance for optimal postoperative pain management in VATS patients.

DETAILED DESCRIPTION:
Video-Assisted Thoracoscopic Surgery (VATS) is a widely used minimally invasive surgical method in thoracic surgery. However, it is known to cause moderate to severe postoperative pain, which can lead to significant respiratory complications such as atelectasis and pneumonia by inhibiting deep breathing and coughing. Inadequate pain control also increases sympathetic nervous system activity, potentially leading to tachycardia, hypertension, and increased myocardial oxygen consumption, especially in patients with cardiac conditions. Furthermore, delayed mobilization due to pain can increase the risk of deep vein thrombosis (DVT) and pulmonary embolism, while insufficient acute pain management may contribute to chronic postoperative pain syndrome. These issues highlight the critical need for effective postoperative pain management. While traditional methods like thoracic epidural analgesia (TEA) and thoracic paravertebral block (TPVB) exist, they are often invasive. In this context, interfascial block techniques such as Edge Laminar Block (ELB) and Serratus Posterior Superior Intercostal Plane Block (SPSIPB) emerge as safer and effective alternatives.

ELB effectively blocks both anterior and posterior branches of thoracic nerves, providing extensive dermatomal sensory loss. It is considered a safer alternative to TPVB due to a lower risk of damage to sensitive structures like the pleura or major vessels during needle placement. ELB has been shown to be effective in postoperative pain management and reducing opioid consumption in surgeries like VATS. SPSIPB, applied by injecting local anesthetic between the serratus posterior superior muscle and intercostal muscles, provides both anteroposterior and lateral thoracic analgesia, creating a broad sensory block area. Studies have reported that SPSIPB provides an effective sensory block between C3-T10 levels and significantly reduces postoperative pain scores.

Study Objectives:

The primary objective of this study is to compare the effectiveness of ELB and SPSIPB in postoperative pain management in patients undergoing VATS. The study will focus on the following specific aims:

To evaluate the effects of ELB and SPSIPB on postoperative pain scores (Visual Analog Scale/Numeric Rating Scale - VAS/NRS).

To compare the potential of both techniques in reducing postoperative opioid consumption.

To examine the incidence of postoperative nausea and vomiting (PONV). To assess secondary outcome measures such as the need for additional analgesics and patient satisfaction in the postoperative period.

This study aims to be one of the first prospective observational studies to directly compare the efficacy of ELB and SPSIPB. The results are expected to provide guidance for optimal postoperative pain management in VATS patients and contribute to a better understanding of the clinical role of these two techniques.

Study Design and Methodology:

This will be a prospective, observational, single-center study. Patient groups will be formed based on natural clinical practice, without randomization. No additional procedures, interventions, or treatment changes will be made to any patient within the scope of the study. All patients will be managed according to standard anesthesia protocols currently applied in the clinic, at the discretion of the responsible anesthesiologists. During the study period, patients undergoing VATS will receive the block protocol routinely preferred by the responsible anesthesiologists, and no intervention will be made by the researchers. This study will not implement a new protocol; rather, it involves prospectively recording data from an anesthesia pain management protocol that proceeds in its natural course.

Postoperative Follow-up:

Pain Assessment: Pain will be assessed using the Visual Analog Scale (VAS) at 1, 4, 12, and 24 hours postoperatively.

Opioid Consumption: The amount of opioid consumed within the first 48 hours will be recorded (as morphine equivalents).

Complications: Complications such as hypotension, pruritus, nausea, and vomiting will be monitored.

Mobilization: The time until first mobilization (sitting at bedside/walking) will be recorded.

Patient Satisfaction: Patient satisfaction and pain control will be monitored and recorded for 48 hours (using a 5-point Likert scale).

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-75 years Scheduled for elective video-assisted thoracoscopic surgery (VATS) American Society of Anesthesiologists (ASA) physical status I-III Ability to provide informed consen

Exclusion Criteria:

Known allergy or contraindication to local anesthetics Chronic opioid use or chronic pain conditions Coagulopathy or use of anticoagulant therapy Infection at the injection site Severe hepatic or renal dysfunction Pregnancy or breastfeeding Inability to understand or complete pain assessment scales

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 18-75 years) scheduled for elective video-assisted thoracoscopic surgery (VATS) at [Your Hospital Name/Institution Name]. These patients will be categorized based on the regional anesthesia technique received (Edge Laminar Block or Serratus Posterior Superior Intercostal Plane Block) for postoperative pain management. Patients with ASA physical status I-III will be included, ensuring a relatively healthy surgical population.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by Visual Analog Scale (VAS) at rest at 2, 6, 12, and 24 hours after surgery. | 2, 6, 12, and 24 hours postoperatively
  Pain intensity will be assessed using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain. The primary outcome is the comparison of VAS scores between the two groups at specified time points.

SECONDARY OUTCOMES:
Total opioid consumption (in mg morphine equivalents) within the first 24 hours after surgery | First 24 hours postoperatively
  The total amount of opioids administered to each patient will be recorded and converted to morphine equivalents for comparison between groups.
Incidence of postoperative complications (e.g., nausea, vomiting, respiratory depression) within 24 hours after surgery. | First 24 hours postoperatively
  The occurrence of common postoperative complications will be documented and compared between groups.
Patient satisfaction with pain management, assessed by a numerical rating scale (1-5) at 24 hours after surgery. | 24 hours postoperatively
  Patients will rate their satisfaction with pain management on a scale from 1 (not satisfied at all) to 5(completely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No